CLINICAL TRIAL: NCT03605524
Title: Olfactory Training and Emotional State
Acronym: ENOLFEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHAO17-WEH/ENOLFEA; 2018-A00653-52 (Other: IdRCB); 2018.05.02 (Other: CPP)
Record Dates: First submitted 2018-07-12; First posted 2018-07-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Depressive Symptoms; Depressive Disorder, Major
Keywords: Sensory training; Depression; Olfaction; Emotion; Perception
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Anosmia | interventions — Smell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensory training (Other): Sensory (Olfactory or visual) training will be done at home for 12 weeks.
  The effect of the training will be evaluated using an experimental protocol includes (i) clinical and psychometric evaluations, (ii) the study of olfactory perception using Sniffin' Sticks Test and (iii) the study of the emotional perception using the "subjective" Sense'n Feel method and the "objective" measurement of the spontaneous pupillary dilatation.
  Interventions: Other: Sensory training

INTERVENTIONS:
Other: Sensory training — 12 weeks sensory training
  Other Names: Olfactory or visual training

SUMMARY:
During the past three decades, researchers have paid particular attention to the study of olfactory disorders in depression. Recent studies have shown that depression is characterized by a change in olfactory and emotional perception resulting in a decrease of the perception of positive stimuli (odors and facial expressions) and an increase in perception of negative stimuli (odors). Moreover, it has also been shown in healthy subjects that the presence of minor depressive symptoms leads to a decreasing of olfactory sensitivity. However, odor discrimination was not impaired in these subjects. This observation suggest the presence of a change in "targeted" olfactory perception in people with depressive symptoms without reporting major depression. In addition, studies in subjects with olfactory disorders (following respiratory tract infections or following Parkinson's disease) have shown an improvement in olfactory function after daily training with odors during 12 weeks.

From all these observations, the hypothesis is that an olfactory training could improve the overall olfactory functioning and the emotional perception of the subjects presenting minor depressive symptoms and of the depressed patients.

DETAILED DESCRIPTION:
Recent studies have shown that depression is characterized by a change in olfactory and emotional perception resulting in a decrease of the perception of positive stimuli (odors and facial expressions) and an increase in perception of negative stimuli (odors). Moreover, it has also been shown in healthy subjects that the presence of minor depressive symptoms leads to a decreasing of olfactory sensitivity. However, odor discrimination was not impaired in these subjects. This observation suggest the presence of a change in "targeted" olfactory perception in people with depressive symptoms without reporting major depression. In addition, studies in subjects with olfactory disorders (following respiratory tract infections or following Parkinson's disease) have shown an improvement in olfactory function after daily training with odors during 12 weeks. Therefore, the hypothesis is that an olfactory training could improve the overall olfactory functioning and the emotional perception of the subjects presenting minor depressive symptoms and of the depressed patients.

The main objective is to study the effect of daily olfactory training on the emotional state and emotional perception of the subject. The effect of the training will be evaluated using three types of evaluations: (1) a clinical evaluation and the psychometric scales, (2) the investigation of the olfactory function and (3) the study of the emotional perception.

The secondary objectives are:

* The identification of olfactory parameters and emotional valences associated with minor depressive symptoms.
* The study of the link between the subjective and objective emotional response on the one hand, and the link between olfactory function, emotional perception and emotional state on the other hand in depressed patients and in individuals with minor depressive symptoms.

ELIGIBILITY:
Inclusion Criteria healthy subjects:

* Without psychiatric history
* QIDS scale score less than or equal to 15
* Affiliation to a social security system
* Able to give his written informed consent

Inclusion Criteria depressed patients:

* With a diagnosis of depressive episode characterized according to the DSM-5 criteria, confirmed by the Mini International Neuropsychiatric Interview (MINI)
* No argument for bipolar disorder or schizophrenia, confirmed by the MINI
* QIDS scale score greater than or equal to 16
* Follow-up in hospitalization and / or ambulatory consultation
* Without comorbidities (alcoholism, eating disorders ...)
* Affiliation to a social security system
* Able to give his written informed consent

Exclusion Criteria healthy subjects and depressed patients:

* Pathology or condition likely to modify their olfactory and / or taste perception
* Allergies with one or more odors, food allergies and / or known anosmias and ageusia
* Legal incapacity and / or circumstances rendering the person incapable of understanding the nature, objectives or consequences of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Olfactory Perception at 3 months | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  Score obtained with the Sniffin 'Stick test

SECONDARY OUTCOMES:
Emotional perception measured Sense'n Feel Method | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  Score obtained with Sense'n Feel Method
Emotional perception measured with SMI RED-m Scientific device | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  Observation of spontaneous pupillary dilatation with SMI RED-m Scientific device
Psychometric scale MINI : Psychiatric disorders exploration | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  Mini International Neuropsychiatric Interview
Psychometric scale TAS-20 : alexithymia assessment | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  Twenty-item toronto Alexithymia Scale (TAS-20)
Psychometric scale STAI-Y : anxiety assessment | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  State Trait Anxiety Inventory
Psychometric scale SHAPS : anhedonia assessment | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  The Snaith-Hamilton Pleasure Scale
Psychometric scale QIDS-SR16 : Depression assessment | Baseline (T0), a month and a half (T1.5), 3 months (T3)
  Quick Inventory of Depressive Symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Wissam EL-HAGE, MD-PhD, Study Director — University Hospital, Tours
Locations (3):
- France (3):
  - University health service, University ,Tours, Tours
  - UMR 1253 IBrain, University, Tours, Tours
  - University Psychiatric Clinic, University hospital,Tours, Tours